CLINICAL TRIAL: NCT03635489
Title: A Phase III Trial of Carboplatin and Paclitaxel Plus Placebo Versus Carboplatin Paclitaxel Plus Concurrent and Extended Bevacizumab in Chinese Women With Newly Diagnosed, Previously Untreated, Stage III or Stage IV Epithelial Ovarian, Fallopian Tube, or Primary Peritoneal Cancer
Brief Title: A Study of the Efficacy and Safety of Bevacizumab in Chinese Women With Newly Diagnosed, Previously Untreated Stage III or Stage IV Epithelial Ovarian, Fallopian Tube, or Primary Peritoneal Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: YO40268
Record Dates: First submitted 2018-08-14; First posted 2018-08-17 (Actual); Results first posted 2023-03-17 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-06

CONDITIONS: Ovarian Cancer; Fallopian Tube Cancer; Primary Peritoneal Cancer
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms | interventions — Paclitaxel; Bevacizumab; Carboplatin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bevacizumab + Paclitaxel + Carboplatin (Experimental): Participants will receive paclitaxel, carboplatin intravenous (IV) infusion on Day 1 of each 21-day cycle for a total of 6 cycles. Bevacizumab IV infusion will start at Cycle 2 for 5 cycles, followed by maintenance therapy up to a maximum of 22 cycles or until disease progression, unacceptable toxicity, or withdrawal, whichever occurs first.
  Interventions: Drug: Paclitaxel; Drug: Bevacizumab; Drug: Carboplatin
- Placebo + Paclitaxel + Carboplatin (Placebo Comparator): Participants will receive paclitaxel, carboplatin IV infusion on Day 1 of each 21-day cycle for a total of 6 cycles. Placebo IV infusion will start at Cycle 2 for 5 cycles, followed by maintenance therapy up to a maximum of 22 cycles or until disease progression, unacceptable toxicity, or withdrawal, whichever occurs first.
  Interventions: Drug: Paclitaxel; Drug: Carboplatin; Drug: Placebo

INTERVENTIONS:
Drug: Paclitaxel — 175 mg/m^2 IV infusion on Day 1 of each 21-day cycle.
Drug: Bevacizumab — 15 mg/kg IV infusion on Day 1 of each 21-day cycle.
  Other Names: Avastin
  Arms: Bevacizumab + Paclitaxel + Carboplatin
Drug: Carboplatin — Area Under the Curve (AUC) of 6 mg/ml/min on Day 1 of each 21-day cycle.
Drug: Placebo — Placebo matched to bevacizumab IV infusion on Day 1 of each 21-day cycle.
  Arms: Placebo + Paclitaxel + Carboplatin

SUMMARY:
This multicenter, double-blind, 2-arm, randomized study will evaluate the efficacy and safety of bevacizumab plus paclitaxel and caboplatin compared with placebo plus paclitaxel and caboplatin in Chinese participants with newly diagnosed, previously untreated Stage III or Stage IV epithelial ovarian, fallopian tube, or primary peritoneal cancer. Participants whose disease has not progressed after six cycles of paclitaxel and carboplatin with either bevacizumab or placebo will continue treatment with either bevacizumab or placebo until disease progression, unacceptable toxicity, or a maximum of 22 cycles, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

* Participants receiving a histologic diagnosis of epithelial ovarian cancer (EOC), peritoneal primary carcinoma, or fallopian tube cancer.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2.
* Life expectancy of at least 12 weeks.
* Adequate hematological, liver, renal and neurologic functions.
* For participants who receive therapeutic anticoagulation: stable anticoagulant regimen.
* Enrollment between 1 and 12 weeks after initial surgery is performed for the combined purpose of diagnosis, staging, and cytoreduction

Exclusion Criteria:

* Current diagnosis of borderline epithelial ovarian tumor or recurrent invasive epithelial ovarian, primary peritoneal, or fallopian tube cancer treated with surgery only.
* Prior radiotherapy to any portion of the abdominal cavity or pelvis.
* Prior chemotherapy for any abdominal or pelvic tumor, including neoadjuvant chemotherapy for ovarian, primary peritoneal, or fallopian tube cancer.
* Any prior targeted therapy (including, but not limited to, vaccines, antibodies, or tyrosine kinase inhibitors) or hormonal therapy for management of their epithelial ovarian or peritoneal primary cancer.
* Synchronous primary endometrial cancer.
* Have a prior history of primary endometrial cancer, except: Stage not greater than Stage IB; no more than superficial myometrial invasion, without vascular or lymphatic invasion; no poorly differentiated subtypes, including papillary serous, clear cell, or other International Federation of Gynecological Oncologists (FIGO) Grade 3 lesions.
* Cancer present within the last 5 years with the exception of non-melanoma-related skin cancers and other specific malignancies or whose previous cancer treatment contraindicates study treatment.
* Active hepatitis B virus (HBV) infection (chronic or acute) or active hepatitis C virus (HCV) infection.
* Serious non-healing wounds, ulcers, or bone fractures.
* Patients with clinically significant cardiovascular disease.
* Have known hypersensitivity to Chinese hamster ovary cell products or other recombinant human or humanized antibodies.
* Have known sensitivity to any component of paclitaxel.
* Undergo major surgical procedure within 28 days prior to randomization or anticipated during the course of the study.
* Have core biopsy or other minor surgical procedures within 7 days prior to the first dose of bevacizumab/placebo.
* History or evidence of thrombotic disorders within the last 6 months prior to enrollment.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-08-15 (Actual); Primary Completion 2021-05-26 (Actual); Study Completion 2023-05-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (16):
- China (16):
  - Beijing Obstetrics and Gynecology Hospital, Capital Medical University, Beijing
  - the First Hospital of Jilin University, Changchun
  - Jilin Cancer Hospital, Changchun
  - Xiangya Hospital Central South University, Changsha
  - West China Second University Hospital, Chengdu
  - Fujian Cancer Hospital, Fuzhou
  - Sun Yet-sen University Cancer Center, Guangzhou
  - Zhejiang Cancer Hospital; Zhejiang Cancer Hospital cancer department, Hangzhou
  - Harbin Medical University Cancer Hospital, Harbin
  - Nanjing Drum Tower Hospital, the Affiliated Hospital of Nanjing University Medical School, Nanjing
  - Guangxi Cancer Hospital of Guangxi Medical University, Nanning
  - Nantong Tumor Hospital, Nantong
  - Fudan University Shanghai Cancer Center, Shanghai
  - Tianjin Medical University General Hospital, Tianjin
  - First Affiliated Hospital of Medical College of Xi'an Jiaotong University, Xi'an
  - Henan Cancer Hospital, Zhengzhou

REFERENCES:
- [Derived] Wu X, Liu J, An R, Yin R, Zhang Y, Zhou H, He A, Wang L, Zhang J, Liu Z, Duan W, Zhu J, Lou G, Chen G, Cheng Y, Xue F, Nick S, Wang H, Li D. First-line bevacizumab plus chemotherapy in Chinese patients with stage III/IV epithelial ovarian cancer, fallopian tube cancer or primary peritoneal cancer: a phase III randomized controlled trial. J Gynecol Oncol. 2024 Sep;35(5):e99. doi: 10.3802/jgo.2024.35.e99. Epub 2024 Apr 22. PMID 38872480
- [Derived] Gaitskell K, Rogozinska E, Platt S, Chen Y, Abd El Aziz M, Tattersall A, Morrison J. Angiogenesis inhibitors for the treatment of epithelial ovarian cancer. Cochrane Database Syst Rev. 2023 Apr 18;4(4):CD007930. doi: 10.1002/14651858.CD007930.pub3. PMID 37185961

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 16 centers in mainland China.
Pre-assignment Details: Participants were randomized with a 1:1 allocation ratio to receive Bevacizumab(B) + Paclitaxel (P) + Carboplatin (C) or Placebo + Paclitaxel + Carboplatin.
Groups:
- Placebo + Paclitaxel + Carboplatin: Participants received paclitaxel, carboplatin intravenous (IV) infusion on Day 1 of each 21-day cycle for a total of 6 cycles. Placebo IV infusion started at Cycle 2 for 5 cycles, followed by maintenance therapy up to a maximum of 22 cycles or until disease progression, unacceptable toxicity, or withdrawal, whichever occurred first.
- Bevacizumab + Paclitaxel + Carboplatin: Participants received paclitaxel, carboplatin IV infusion on Day 1 of each 21-day cycle for a total of 6 cycles. Bevacizumab IV infusion started at Cycle 2 for 5 cycles, followed by maintenance therapy up to a maximum of 22 cycles or until disease progression, unacceptable toxicity, or withdrawal, whichever occurred first.
Period: Overall Study
Arm/Group | Placebo + Paclitaxel + Carboplatin | Bevacizumab + Paclitaxel + Carboplatin
Started | 49 | 51
Completed | 0 | 0
Not Completed | 49 | 51
Not completed — Death | 19 | 13
Not completed — Lost to Follow-up | 1 | 2
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Study Ended by Sponsor | 28 | 34

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo + Paclitaxel + Carboplatin | Bevacizumab + Paclitaxel + Carboplatin | Total
Number analyzed (Participants) | 49 | 51 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.1 (8.4) | 54.1 (8.2) | 53.6 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49 | 51 | 100
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 49 | 51 | 100
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 49 | 51 | 100
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS)
Description: PFS was defined as time from randomization to the first occurrence of disease progression, as assessed by the Investigator using RECIST v1.1, or death from any cause, whichever occurs first.
Time Frame: Randomization up to disease progression or death from any cause, whichever occurs first (up to approximately 24 months)
Population: The intent-to-treat (ITT) population was defined as all randomized participants regardless of whether the assigned study treatment was received. For efficacy analyses, participants were analyzed according to their randomized treatment assignment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo + Paclitaxel + Carboplatin | Bevacizumab + Paclitaxel + Carboplatin
Number analyzed (Participants) | 49 | 51
months | 12.32 [9.53 to 15.05] | 22.57 [18.60 to NA] — The upper bound of the 95% confidence interval (CI) was not reached.
Statistical Analysis 1: Comparison: Placebo + Paclitaxel + Carboplatin vs Bevacizumab + Paclitaxel + Carboplatin; Test type: Superiority — Stratified Analysis; p < .0001, Regression, Cox; Hazard Ratio (HR) = 0.30, 95% CI 2-sided [0.17 to 0.53]
Statistical Analysis 2: Comparison: Placebo + Paclitaxel + Carboplatin vs Bevacizumab + Paclitaxel + Carboplatin; Test type: Superiority — Unstratified Analysis; p < .0001, Regression, Cox; Hazard Ratio (HR) = 0.34, 95% CI 2-sided [0.20 to 0.58]

2. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from the date of randomization to the date of death from any cause.
Time Frame: Randomization up to to death from any cause (up to approximately 54.1 months)
Population: The ITT population was defined as all randomized participants regardless of whether the assigned study treatment was received. For efficacy analyses, participants were analyzed according to their randomized treatment assignment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo + Paclitaxel + Carboplatin | Bevacizumab + Paclitaxel + Carboplatin
Number analyzed (Participants) | 49 | 51
months | 48.89 [40.31 to NA] — Insufficient number of participants with events. | NA [NA to NA] — Insufficient number of participants with events.
Statistical Analysis 1: Comparison: Placebo + Paclitaxel + Carboplatin vs Bevacizumab + Paclitaxel + Carboplatin; Test type: Superiority — Unstratified analysis; Hazard Ratio (HR) = 0.60, 95% CI 2-sided [0.30 to 1.21]

3. Secondary Outcome: Objective Response Rate (ORR)
Description: ORR was defined as the proportion of participants with complete response (CR) or partial response (PR) as assessed by investigator according to RECIST v.1.1.
Time Frame: Randomization up to disease progression or death from any cause, whichever occurs first (up to approximately 24 months)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo + Paclitaxel + Carboplatin | Bevacizumab + Paclitaxel + Carboplatin
Number analyzed (Participants) | 28 | 24
percentage of participants | 92.9 [76.50 to 99.12] | 95.8 [78.88 to 99.89]

4. Secondary Outcome: Duration of Response (DOR)
Description: DOR was defined as the time from when response (CR or PR) was first documented to first documented disease progression,as assessed by the Investigator using RECIST v1.1, or death from any cause, whichever occurred first. DOR was evaluated for participants who had a objective response of CR or PR.
Time Frame: From the date of first occurrence of a complete or partial response until disease progression or death from any cause (up to approximately 24 months)
Population: The intent-to-treat (ITT) population was defined as all randomized participants regardless of whether the assigned study treatment was received. Here, all randomized participants who had an objective response (CR or PR) by the investigator per RECIST v1.1 were included in the analysis.
Measure: Median (80% Confidence Interval); unit: months
Arm/Group | Placebo + Paclitaxel + Carboplatin | Bevacizumab + Paclitaxel + Carboplatin
Number analyzed (Participants) | 26 | 23
months | 8.87 [7.56 to 13.14] | 16.10 [10.81 to NA] — The upper bound of 95% CI was not reached

5. Secondary Outcome: Percentage of Participants Who Report a Clinically Meaningful Improvement in Patient-Reported Abdominal Pain
Description: A clinically meaningful improvement in patient-reported abdominal pain or bloating was defined as a ≥10-point decrease from the linearly transformed 0-100 point baseline symptom scale score on each of two items from the Abdominal/Gastrointestinal Symptom Scale of the European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire - Ovarian Cancer Module (QLQ-OV28).
Time Frame: From randomization to the end of treatment/discontinuation (up to approximately 70 weeks), and during follow-up period (up to approximately 24 months)
Population: The intent-to-treat (ITT) population was defined as all randomized participants regardless of whether the assigned study treatment was received. Here, all randomized participants who had a baseline and ≥1 post-baseline PRO assessment were included in the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo + Paclitaxel + Carboplatin | Bevacizumab + Paclitaxel + Carboplatin
Number analyzed (Participants) | 48 | 50
percentage of participants
  Cycle 4 Day 1: number analyzed (Participants) | 46 | 48
  Cycle 4 Day 1 | 37.0 [23.21 to 52.45] | 31.3 [18.66 to 46.25]
  Cycle 7 Day 1: number analyzed (Participants) | 44 | 38
  Cycle 7 Day 1 | 40.9 [26.34 to 56.75] | 42.1 [26.31 to 58.18]
  Cycle 13 Day 1: number analyzed (Participants) | 31 | 35
  Cycle 13 Day 1 | 48.4 [30.15 to 66.94] | 40.0 [23.87 to 57.89]
  Cycle 22 Day 1: number analyzed (Participants) | 16 | 25
  Cycle 22 Day 1 | 37.5 [15.20 to 64.57] | 48.0 [27.80 to 68.69]
  Treatment Completion / Early Termination Visit: number analyzed (Participants) | 45 | 42
  Treatment Completion / Early Termination Visit | 37.8 [23.77 to 53.46] | 45.2 [29.85 to 61.33]
  Survival Follow Up 3 Months: number analyzed (Participants) | 27 | 36
  Survival Follow Up 3 Months | 37.0 [19.40 to 57.63] | 33.3 [18.56 to 50.97]
  Survival Follow Up 6 Months: number analyzed (Participants) | 15 | 21
  Survival Follow Up 6 Months | 33.3 [11.82 to 61.62] | 38.1 [18.11 to 61.56]
  Survival Follow Up 9 Months: number analyzed (Participants) | 8 | 13
  Survival Follow Up 9 Months | 50.0 [15.70 to 84.30] | 46.2 [19.22 to 74.87]
  Survival Follow Up 12 Months: number analyzed (Participants) | 7 | 7
  Survival Follow Up 12 Months | 14.3 [0.36 to 57.87] | 42.9 [9.90 to 81.59]
  Survival Follow Up 18 Months: number analyzed (Participants) | 0 | 3
  Survival Follow Up 18 Months |  | 66.7 [9.43 to 99.16]
  Survival Follow Up 24 Months: number analyzed (Participants) | 0 | 1
  Survival Follow Up 24 Months |  | 0 [0 to 97.50]

6. Secondary Outcome: Percentage of Participants Who Report a Clinically Meaningful Improvement in Patient-Reported Bloating
Description: as for outcome 5
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo + Paclitaxel + Carboplatin | Bevacizumab + Paclitaxel + Carboplatin
Number analyzed (Participants) | 48 | 50
percentage of participants
  Cycle 4 Day 1: number analyzed (Participants) | 46 | 48
  Cycle 4 Day 1 | 26.1 [14.27 to 41.13] | 33.3 [20.40 to 48.41]
  Cycle 7 Day 1: number analyzed (Participants) | 44 | 38
  Cycle 7 Day 1 | 36.4 [22.41 to 52.23] | 47.4 [30.98 to 64.18]
  Cycle 13 Day 1: number analyzed (Participants) | 31 | 35
  Cycle 13 Day 1 | 29.0 [14.22 to 48.04] | 31.4 [16.85 to 49.29]
  Cycle 22 Day 1: number analyzed (Participants) | 16 | 25
  Cycle 22 Day 1 | 25.0 [7.27 to 52.38] | 40.0 [21.13 to 61.33]
  Treatment Completion / Early Termination Visit: number analyzed (Participants) | 45 | 42
  Treatment Completion / Early Termination Visit | 33.3 [20.00 to 48.95] | 33.3 [19.57 to 49.55]
  Survival Follow Up 3 Months: number analyzed (Participants) | 27 | 36
  Survival Follow Up 3 Months | 25.9 [11.11 to 46.28] | 33.3 [18.56 to 50.97]
  Survival Follow Up 6 Months: number analyzed (Participants) | 15 | 21
  Survival Follow Up 6 Months | 46.7 [21.27 to 73.41] | 19.0 [5.45 to 41.91]
  Survival Follow Up 9 Months: number analyzed (Participants) | 8 | 13
  Survival Follow Up 9 Months | 25.0 [3.19 to 65.09] | 23.1 [5.04 to 53.81]
  Survival Follow Up 12 Months: number analyzed (Participants) | 7 | 7
  Survival Follow Up 12 Months | 28.6 [3.67 to 70.96] | 28.6 [3.67 to 70.96]
  Survival Follow Up 18 Months: number analyzed (Participants) | 0 | 3
  Survival Follow Up 18 Months |  | 66.7 [9.43 to 99.16]
  Survival Follow Up 24 Months: number analyzed (Participants) | 0 | 1
  Survival Follow Up 24 Months |  | 0 [0 to 97.50]

7. Secondary Outcome: Percentage of Participants Who Report a Clinically Meaningful Improvement in Patient-Reported Function (Physical)
Description: A clinically meaningful improvement in patient-reported function and HRQoL was defined as a >10-point increase from the linearly transformed 0-100 point baseline scale score on each of the four functional (physical, role, emotional, social) scales and global health status/HRQoL scale of the European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire - Core 30 (QLQ-C30).
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo + Paclitaxel + Carboplatin | Bevacizumab + Paclitaxel + Carboplatin
Number analyzed (Participants) | 48 | 50
percentage of participants
  Cycle 4 Day 1: number analyzed (Participants) | 46 | 48
  Cycle 4 Day 1 | 17.4 [7.82 to 31.42] | 16.7 [7.48 to 30.22]
  Cycle 7 Day 1: number analyzed (Participants) | 44 | 38
  Cycle 7 Day 1 | 18.2 [8.19 to 32.71] | 18.4 [7.74 to 34.33]
  Cycle 13 Day 1: number analyzed (Participants) | 31 | 35
  Cycle 13 Day 1 | 45.2 [27.32 to 63.97] | 34.3 [19.13 to 52.21]
  Cycle 22 Day 1: number analyzed (Participants) | 16 | 25
  Cycle 22 Day 1 | 43.8 [19.75 to 70.12] | 36.0 [17.97 to 57.48]
  Treatment Completion / Early Termination Visit: number analyzed (Participants) | 45 | 42
  Treatment Completion / Early Termination Visit | 31.1 [18.17 to 46.65] | 31.0 [17.62 to 47.09]
  Survival Follow Up 3 Months: number analyzed (Participants) | 27 | 36
  Survival Follow Up 3 Months | 44.4 [25.48 to 64.67] | 27.8 [14.20 to 45.19]
  Survival Follow Up 6 Months: number analyzed (Participants) | 15 | 21
  Survival Follow Up 6 Months | 13.3 [1.66 to 40.46] | 23.8 [8.22 to 47.17]
  Survival Follow Up 9 Months: number analyzed (Participants) | 8 | 13
  Survival Follow Up 9 Months | 12.5 [0.32 to 52.65] | 23.1 [5.04 to 53.81]
  Survival Follow Up 12 Months: number analyzed (Participants) | 7 | 7
  Survival Follow Up 12 Months | 14.3 [0.36 to 57.87] | 28.6 [3.67 to 70.96]
  Survival Follow Up 18 Months: number analyzed (Participants) | 0 | 3
  Survival Follow Up 18 Months |  | 0 [0 to 70.76]
  Survival Follow Up 24 Months: number analyzed (Participants) | 0 | 1
  Survival Follow Up 24 Months |  | 0 [0 to 97.50]

8. Secondary Outcome: Percentage of Participants Who Report a Clinically Meaningful Improvement in Patient-Reported Function (Role)
Description: as for outcome 7
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo + Paclitaxel + Carboplatin | Bevacizumab + Paclitaxel + Carboplatin
Number analyzed (Participants) | 48 | 50
percentage of participants
  Cycle 4 Day 1: number analyzed (Participants) | 46 | 48
  Cycle 4 Day 1 | 34.8 [21.35 to 50.25] | 31.3 [18.66 to 46.25]
  Cycle 7 Day 1: number analyzed (Participants) | 44 | 38
  Cycle 7 Day 1 | 25.0 [13.19 to 40.34] | 36.8 [21.81 to 54.01]
  Cycle 13 Day 1: number analyzed (Participants) | 31 | 35
  Cycle 13 Day 1 | 45.2 [27.32 to 63.97] | 48.6 [31.38 to 66.01]
  Cycle 22 Day 1: number analyzed (Participants) | 16 | 25
  Cycle 22 Day 1 | 50.0 [24.65 to 75.35] | 40.0 [21.13 to 61.33]
  Treatment Completion / Early Termination Visit: number analyzed (Participants) | 45 | 42
  Treatment Completion / Early Termination Visit | 40.0 [25.70 to 55.67] | 42.9 [27.72 to 59.04]
  Survival Follow Up 3 Months: number analyzed (Participants) | 27 | 36
  Survival Follow Up 3 Months | 48.1 [28.67 to 68.05] | 33.3 [18.56 to 50.97]
  Survival Follow Up 6 Months: number analyzed (Participants) | 15 | 21
  Survival Follow Up 6 Months | 40.0 [16.34 to 67.71] | 42.9 [21.82 to 65.98]
  Survival Follow Up 9 Months: number analyzed (Participants) | 8 | 13
  Survival Follow Up 9 Months | 37.5 [8.52 to 75.51] | 30.8 [9.09 to 61.43]
  Survival Follow Up 12 Months: number analyzed (Participants) | 7 | 7
  Survival Follow Up 12 Months | 42.9 [9.90 to 81.59] | 57.1 [18.41 to 90.10]
  Survival Follow Up 18 Months: number analyzed (Participants) | 0 | 3
  Survival Follow Up 18 Months |  | 33.3 [0.84 to 90.57]
  Survival Follow Up 24 Months: number analyzed (Participants) | 0 | 1
  Survival Follow Up 24 Months |  | 0 [0 to 97.50]

9. Secondary Outcome: Percentage of Participants Who Report a Clinically Meaningful Improvement in Patient-Reported Function (Social)
Description: as for outcome 7
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo + Paclitaxel + Carboplatin | Bevacizumab + Paclitaxel + Carboplatin
Number analyzed (Participants) | 48 | 50
percentage of participants
  Cycle 4 Day 1: number analyzed (Participants) | 46 | 48
  Cycle 4 Day 1 | 28.3 [15.99 to 43.46] | 29.2 [16.95 to 44.06]
  Cycle 7 Day 1: number analyzed (Participants) | 44 | 38
  Cycle 7 Day 1 | 27.3 [14.96 to 42.79] | 28.9 [15.42 to 45.90]
  Cycle 13 Day 1: number analyzed (Participants) | 31 | 35
  Cycle 13 Day 1 | 38.7 [21.85 to 57.81] | 28.6 [14.64 to 46.30]
  Cycle 22 Day 1: number analyzed (Participants) | 16 | 25
  Cycle 22 Day 1 | 43.8 [19.75 to 70.12] | 36.0 [17.97 to 57.48]
  Treatment Completion / Early Termination Visit: number analyzed (Participants) | 45 | 42
  Treatment Completion / Early Termination Visit | 28.9 [16.37 to 44.31] | 33.3 [19.57 to 49.55]
  Survival Follow Up 3 Months: number analyzed (Participants) | 27 | 36
  Survival Follow Up 3 Months | 33.3 [16.52 to 53.96] | 47.2 [30.41 to 64.51]
  Survival Follow Up 6 Months: number analyzed (Participants) | 15 | 21
  Survival Follow Up 6 Months | 26.7 [7.79 to 55.10] | 28.6 [11.28 to 52.18]
  Survival Follow Up 9 Months: number analyzed (Participants) | 8 | 13
  Survival Follow Up 9 Months | 37.5 [8.52 to 75.51] | 7.7 [0.19 to 36.03]
  Survival Follow Up 12 Months: number analyzed (Participants) | 7 | 7
  Survival Follow Up 12 Months | 28.6 [3.67 to 70.96] | 28.6 [3.67 to 70.96]
  Survival Follow Up 18 Months: number analyzed (Participants) | 0 | 3
  Survival Follow Up 18 Months |  | 66.7 [9.43 to 99.16]
  Survival Follow Up 24 Months: number analyzed (Participants) | 0 | 1
  Survival Follow Up 24 Months |  | 100 [2.50 to 100]

10. Secondary Outcome: Percentage of Participants Who Report a Clinically Meaningful Improvement in Patient-Reported Function (Emotional)
Description: as for outcome 7
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo + Paclitaxel + Carboplatin | Bevacizumab + Paclitaxel + Carboplatin
Number analyzed (Participants) | 48 | 50
percentage of participants
  Cycle 4 Day 1: number analyzed (Participants) | 46 | 48
  Cycle 4 Day 1 | 8.7 [2.42 to 20.79] | 22.9 [12.03 to 37.31]
  Cycle 7 Day 1: number analyzed (Participants) | 44 | 38
  Cycle 7 Day 1 | 13.6 [5.17 to 27.35] | 21.1 [9.55 to 37.32]
  Cycle 13 Day 1: number analyzed (Participants) | 31 | 35
  Cycle 13 Day 1 | 9.7 [2.04 to 25.75] | 25.7 [12.49 to 43.26]
  Cycle 22 Day 1: number analyzed (Participants) | 16 | 25
  Cycle 22 Day 1 | 18.8 [4.05 to 45.65] | 28.0 [12.07 to 49.39]
  Treatment Completion / Early Termination Visit: number analyzed (Participants) | 45 | 42
  Treatment Completion / Early Termination Visit | 11.1 [3.71 to 24.05] | 21.4 [10.30 to 36.81]
  Survival Follow Up 3 Months: number analyzed (Participants) | 27 | 36
  Survival Follow Up 3 Months | 22.2 [8.62 to 42.26] | 27.8 [14.20 to 45.19]
  Survival Follow Up 6 Months: number analyzed (Participants) | 15 | 21
  Survival Follow Up 6 Months | 6.7 [0.17 to 31.95] | 38.1 [18.11 to 61.56]
  Survival Follow Up 9 Months: number analyzed (Participants) | 8 | 13
  Survival Follow Up 9 Months | 12.5 [0.32 to 57.87] | 38.5 [13.86 to 68.42]
  Survival Follow Up 12 Months: number analyzed (Participants) | 7 | 7
  Survival Follow Up 12 Months | 14.3 [0.36 to 57.87] | 28.6 [3.67 to 70.96]
  Survival Follow Up 18 Months: number analyzed (Participants) | 0 | 3
  Survival Follow Up 18 Months |  | 0 [0 to 70.76]
  Survival Follow Up 24 Months: number analyzed (Participants) | 0 | 1
  Survival Follow Up 24 Months |  | 0 [0 to 97.50]

11. Secondary Outcome: Pecentage of Participants Who Report a Clinically Meaningful Improvement in Patient-Reported Health Related Quality of Life (HRQoL)
Description: as for outcome 7
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo + Paclitaxel + Carboplatin | Bevacizumab + Paclitaxel + Carboplatin
Number analyzed (Participants) | 48 | 50
percentage of participants
  Cycle 4 Day 1: number analyzed (Participants) | 46 | 48
  Cycle 4 Day 1 | 19.6 [9.36 to 33.91] | 33.3 [20.40 to 48.41]
  Cycle 7 Day 1: number analyzed (Participants) | 44 | 38
  Cycle 7 Day 1 | 34.1 [20.49 to 49.92] | 34.2 [19.63 to 51.35]
  Cycle 13 Day 1: number analyzed (Participants) | 31 | 35
  Cycle 13 Day 1 | 38.7 [21.85 to 57.81] | 34.3 [19.13 to 52.21]
  Cycle 22 Day 1: number analyzed (Participants) | 16 | 25
  Cycle 22 Day 1 | 43.8 [19.75 to 70.12] | 44.0 [24.40 to 65.07]
  Treatment Completion / Early Termination Visit: number analyzed (Participants) | 45 | 42
  Treatment Completion / Early Termination Visit | 31.1 [18.17 to 46.65] | 40.5 [25.63 to 56.72]
  Survival Follow Up 3 Months: number analyzed (Participants) | 27 | 36
  Survival Follow Up 3 Months | 29.6 [13.75 to 50.18] | 38.9 [23.14 to 56.54]
  Survival Follow Up 6 Months: number analyzed (Participants) | 15 | 21
  Survival Follow Up 6 Months | 33.3 [11.82 to 61.62] | 28.6 [11.28 to 52.18]
  Survival Follow Up 9 Months: number analyzed (Participants) | 8 | 13
  Survival Follow Up 9 Months | 12.5 [0.32 to 52.65] | 23.1 [5.04 to 53.81]
  Survival Follow Up 12 Months: number analyzed (Participants) | 7 | 7
  Survival Follow Up 12 Months | 14.3 [0.36 to 57.87] | 42.9 [9.90 to 81.59]
  Survival Follow Up 18 Months: number analyzed (Participants) | 0 | 3
  Survival Follow Up 18 Months |  | 33.3 [0.84 to 90.57]
  Survival Follow Up 24 Months: number analyzed (Participants) | 0 | 1
  Survival Follow Up 24 Months |  | 0 [0 to 97.50]

12. Secondary Outcome: Percentage of Participants With Adverse Events (AEs)
Time Frame: From randomization up to 90 days after last dose of study treatment or until initiation of new anti-cancer therapy (up to approximately 76 weeks)
Population: The safety population was defined as participants who received any amount of any component of the study treatments (bevacizumab, paclitaxel or carboplatin). Participants were allocated to treatment arms according to the treatment they actually received (i.e., participants randomized to placebo + chemotherapy alone who received at least one full or partial dose of bevacizumab were included in the bevacizumab + chemotherapy arm for safety).
Measure: Number; unit: percentage of participants
Arm/Group | Placebo + Paclitaxel + Carboplatin | Bevacizumab + Paclitaxel + Carboplatin
Number analyzed (Participants) | 50 | 49
percentage of participants | 100 | 100

ADVERSE EVENTS:
Time Frame: All-cause mortality: From randomization up to end of follow up (54.1 months) AEs and SAEs: From randomization up to 90 days after last dose of study treatment or until initiation of new anti-cancer therapy (up to approximately 76 weeks)
Description: Safety population: participants who received any amount of study treatment (Bev,C or P). Participants were allocated to treatment arms per actual treatment received. 1 participant in Bev+P+C arm withdrew before receiving treatment & was excluded from safety population. 2 participants in Bev+P+C arm did not receive Bev, & were included in Placebo+P+C arm in safety population. 1 participant in Placebo+P+C arm received partial bevacizumab dose & was included in B+P+C arm in safety population.
Arm/Group | Placebo + Paclitaxel + Carboplatin | Bevacizumab + Paclitaxel + Carboplatin
All-Cause Mortality (participants affected / at risk) | 19/50 | 13/49
Serious Adverse Events (participants affected / at risk) | 16/50 | 17/49
Other Adverse Events (participants affected / at risk) | 49/50 | 49/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo + Paclitaxel + Carboplatin (N=50) | Bevacizumab + Paclitaxel + Carboplatin (N=49)
Anaemia (Blood and lymphatic system disorders) | 3 (5) | 0 (0)
Granulocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Myelosuppression (Blood and lymphatic system disorders) | 5 (6) | 4 (6)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0)
Femoral hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 2 (2)
Intestinal obstruction (Gastrointestinal disorders) | 2 (2) | 2 (2)
Mechanical ileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 1 (1)
Subileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 1 (1)
Anaphylactic shock (Immune system disorders) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 1 (1)
Granulocyte count decreased (Investigations) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 3 (3) | 0 (0)
Platelet count decreased (Investigations) | 5 (9) | 3 (3)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Pelvic haematoma (Reproductive system and breast disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo + Paclitaxel + Carboplatin (N=50) | Bevacizumab + Paclitaxel + Carboplatin (N=49)
Anaemia (Blood and lymphatic system disorders) | 35 (118) | 38 (101)
Leukopenia (Blood and lymphatic system disorders) | 14 (72) | 12 (47)
Myelosuppression (Blood and lymphatic system disorders) | 5 (7) | 6 (16)
Neutropenia (Blood and lymphatic system disorders) | 7 (20) | 6 (15)
Thrombocytopenia (Blood and lymphatic system disorders) | 6 (25) | 6 (15)
Sinus arrhythmia (Cardiac disorders) | 1 (4) | 4 (10)
Sinus bradycardia (Cardiac disorders) | 2 (3) | 3 (6)
Sinus tachycardia (Cardiac disorders) | 2 (2) | 3 (4)
Abdominal distension (Gastrointestinal disorders) | 5 (6) | 3 (4)
Abdominal pain (Gastrointestinal disorders) | 11 (15) | 10 (15)
Abdominal pain lower (Gastrointestinal disorders) | 3 (4) | 3 (4)
Abdominal pain upper (Gastrointestinal disorders) | 5 (7) | 3 (3)
Constipation (Gastrointestinal disorders) | 10 (26) | 15 (24)
Diarrhoea (Gastrointestinal disorders) | 9 (12) | 6 (10)
Flatulence (Gastrointestinal disorders) | 3 (3) | 1 (1)
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 4 (5)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 3 (4)
Nausea (Gastrointestinal disorders) | 25 (62) | 20 (41)
Toothache (Gastrointestinal disorders) | 0 (0) | 5 (8)
Vomiting (Gastrointestinal disorders) | 21 (51) | 13 (25)
Asthenia (General disorders) | 6 (9) | 3 (8)
Chest discomfort (General disorders) | 3 (3) | 2 (2)
Fatigue (General disorders) | 2 (4) | 7 (7)
Influenza like illness (General disorders) | 5 (7) | 5 (7)
Malaise (General disorders) | 6 (21) | 12 (25)
Oedema peripheral (General disorders) | 2 (3) | 3 (3)
Pain (General disorders) | 12 (21) | 5 (11)
Pyrexia (General disorders) | 3 (3) | 2 (2)
Hepatic function abnormal (Hepatobiliary disorders) | 7 (13) | 7 (9)
Pharyngitis (Infections and infestations) | 0 (0) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 6 (11) | 9 (17)
Urinary tract infection (Infections and infestations) | 1 (2) | 6 (7)
Alanine aminotransferase increased (Investigations) | 19 (48) | 17 (36)
Aspartate aminotransferase increased (Investigations) | 14 (32) | 13 (39)
Blood alkaline phosphatase increased (Investigations) | 4 (9) | 8 (20)
Blood bilirubin increased (Investigations) | 2 (4) | 4 (10)
Blood glucose increased (Investigations) | 3 (4) | 1 (1)
Blood lactate dehydrogenase increased (Investigations) | 3 (10) | 4 (11)
Blood urea increased (Investigations) | 2 (2) | 6 (14)
Electrocardiogram T wave abnormal (Investigations) | 1 (3) | 5 (21)
Gamma-glutamyltransferase increased (Investigations) | 5 (11) | 10 (26)
Neutrophil count decreased (Investigations) | 32 (227) | 39 (250)
Platelet count decreased (Investigations) | 26 (83) | 29 (88)
Protein urine present (Investigations) | 2 (5) | 7 (9)
Red blood cells urine positive (Investigations) | 3 (3) | 1 (1)
Urinary occult blood positive (Investigations) | 5 (9) | 0 (0)
Weight decreased (Investigations) | 5 (8) | 4 (4)
Weight increased (Investigations) | 11 (11) | 7 (7)
White blood cell count decreased (Investigations) | 29 (186) | 38 (226)
White blood cells urine positive (Investigations) | 5 (6) | 8 (11)
Decreased appetite (Metabolism and nutrition disorders) | 7 (7) | 14 (28)
Dyslipidaemia (Metabolism and nutrition disorders) | 0 (0) | 4 (4)
Hyperglycaemia (Metabolism and nutrition disorders) | 7 (13) | 10 (17)
Hyperuricaemia (Metabolism and nutrition disorders) | 3 (6) | 7 (11)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 5 (10) | 1 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 8 (15) | 8 (11)
Hypoproteinaemia (Metabolism and nutrition disorders) | 3 (3) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 (15) | 6 (6)
Bone pain (Musculoskeletal and connective tissue disorders) | 3 (8) | 2 (6)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3 (4) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (6) | 4 (6)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 (16) | 11 (15)
Dizziness (Nervous system disorders) | 7 (9) | 4 (4)
Hypoaesthesia (Nervous system disorders) | 17 (20) | 17 (24)
Memory impairment (Nervous system disorders) | 4 (4) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 6 (10) | 11 (13)
Insomnia (Psychiatric disorders) | 8 (13) | 10 (23)
Haematuria (Renal and urinary disorders) | 2 (2) | 4 (4)
Leukocyturia (Renal and urinary disorders) | 2 (2) | 3 (7)
Proteinuria (Renal and urinary disorders) | 3 (4) | 22 (41)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 6 (6)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (4)
Alopecia (Skin and subcutaneous tissue disorders) | 41 (43) | 43 (43)
Night sweats (Skin and subcutaneous tissue disorders) | 3 (3) | 3 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 7 (9) | 5 (6)
Hypertension (Vascular disorders) | 9 (16) | 18 (65)
Neuropathy peripheral (Nervous system disorders) | 4 (4) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2019-11-04): https://cdn.clinicaltrials.gov/large-docs/89/NCT03635489/Prot_000.pdf
  • Statistical Analysis Plan (2020-12-04): https://cdn.clinicaltrials.gov/large-docs/89/NCT03635489/SAP_001.pdf